CLINICAL TRIAL: NCT05158855
Title: Human Pilot Test of an Oral Neutralizing Antibody Booster for Post-vaccinated People With COVID19 Vaccine
Brief Title: Oral Neutralizing Antibody Booster for Post-vaccinated People With COVID19 Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DreamTec Research Limited (Industry)
Collaborators: DreamTec Cytokine Limited (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRP/008/21FXBooster
Record Dates: First submitted 2021-12-14; First posted 2021-12-15 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Volunteers who vaccinated with COVID-19 vaccines for over 6 months will be recruited and will receive 1 capsule of neutralizing antibody booster. Their weight, blood pressure, and the concentration of neutralizing IgG antibody against receptor binding domain of spike protein in SARS-CoV2 will be measured before the oral administration and 14, 28 days after the administration. Number of adverse event from the beginning of the administration to 30 days after the administration will also be recorded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neutralizing antibody booster for vaccinated participants (Experimental): participants after 6-month vaccinated with COVID-19 vaccine received 1 capsule of B. subtilis spore extract
  Interventions: Dietary Supplement: Bacillus subtilis spore extract

INTERVENTIONS:
Dietary Supplement: Bacillus subtilis spore extract — Bacillus subtilis, a harmless intestinal commensal, has earned in recent years, great reputation as a vaccine production host and delivery vector with advantages such as low cost, safe for human consumption and straightforward administration. The technology team has succeeded engineering Bacillus subtilis with spore coat proteins resembling the proteins of the nucleus and spikes of coronavirus. This product could have a vaccine like activity within the intestinal environment.

SUMMARY:
This is a study trial to assess the effectiveness of the immune response stimulated by the genetically engineered Bacillus subtilis spore extract which contain Spike protein of the SARS-COV2 on the spore coat.

DETAILED DESCRIPTION:
COVID-19 immunization reduces the risk of COVID-19 and potentially serious complications. In clinical trials, all COVID-19 vaccines currently authorized for use in the United States are beneficial in protecting adults and children 5 years and older against COVID-19, including severe illness. So far, studies looking at how COVID-19 vaccines work in real-world conditions (vaccine effectiveness studies) have shown that they work well. However, it has been reported that most of the antibodies in people who received the second dose of COVID-19 vaccine had been dramatically decreased.

Bacillus subtilis (B. subtilis) is a generally regarded as safe organism and it is a common food source. The investigators have used an engineered Bacillus subtilis spore which express and display the spike protein receptor binding domain (sRBD) of the SARS-CoV-2 on the surface. The investigators have proved that it successfully increased the neutralizing antibody against sRBD in unvaccinated mice and human individuals after oral administration.

On this basis, the investigators designed and developed an oral antibody booster by extracting the spore surface of B. subtilis. This supplement has the advantage of being stable and effective, free of recombinant plasmid, and can be served as a potential antibody booster to existing vaccines.

Mice toxicity and efficacy test was conducted and the experiment proved that the B. subtilis spores extract was effective in inducing immune response, and it was safe and did not cause any significant adverse effect.

The B. subtilis spore extract will be further studied in a human trials through oral administration to test its safety and the immune effect resulted in human body.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* age over 12 years
* the outcome of the following examinations should be clinically insignificant: medical and surgical history (hypo-, hypertension, allergy, other diseases, major surgery, micturition, defecation, sleep, illness within the last 4 weeks prior to the start of the trial);
* participant vaccinated with COVID-19 over 6 months
* anti-SARS CoV 2 neutralizing antibody is negative in serum.

Exclusion Criteria:

* pregnant women
* history of COVID-19 infection or showing COVID-19 infection symptoms
* having had contact to people with known COVID-19 infection in the last 14 days
* having fever (> 37.4oC in the last 24 hours), dry cough or feeling tired and having aches and pains, nasal congestion, runny nose, sore throat and diarrhea.
* positive real time RT-PCR COVID-19 test.
* persons with autoimmune diseases
* allergic diathesis or any clinically significant allergic disease (i.e. asthma)
* any condition that might impair the immune response
* recent or current immunosuppressive medication
* any other vaccine application 5 months before the first dose

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
To assess the safety of the engineered Bacillus subtilis spore coat extract | 3 months
  To measure the weight changes in kilograms and number of incidence of adverse event from the beginning of the administration to 30 days after the administration
Concentration of Neutralizing IgG antibody against Receptor binding domain of spike protein of SARS-CoV2 | 3 months
  To measure the concentration of Neutralizing IgG antibody against Receptor binding domain of spike protein of SARS-CoV2 before the administration and 14, 28 days after the administration

CONTACTS AND LOCATIONS:
Overall Officials: WAI YEUNG KWONG, PhD, Study Director — DreamTec Cytokine Limited
Locations (1):
- Macao Greater Bay Area Association of Healthcare Providers, Macao, Macau

IPD SHARING:
Plan to Share IPD: No